CLINICAL TRIAL: NCT00216736
Title: Does a Single Oral Dose of Dexamethasone After Successful Emergency Treatment of Migraine Reduce the Incidence or Severity of Rebound Headache Within 48 Hours?
Brief Title: Oral Dexamethasone for Treatment of Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Joseph Epstein Centre for Emergency Medicine Research (Other)
Responsible Party: Principal Investigator, Professor Anne-Maree Kelly, Director JECEMR, The Joseph Epstein Centre for Emergency Medicine Research
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2004.221
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Migraine
Keywords: Migraine; Headache; Rebound headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): This group received intravenous phenothiazine treatment for migraine (dosing at physician discretion) plus placebo. Patients and clinicians were blinded.
  Interventions: Drug: placebo
- 2 (Experimental): This group received intravenous phenothiazine migraine treatment (dosage at physician discretion) plus oral dexamethasone 8mg at time of emergency department discharge. Patients and clinicians were blinded.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Single dose oral dexamethasone 8mg at time of ED discharge
  Arms: 2
Drug: placebo — Single dose oral placebo at ED discharge
  Arms: 1

SUMMARY:
The aim of this project is to determine if a single dose of oral dexamethasone at the time of discharge from the emergency department (ED) [after successful treatment] prevents rebound headache.

Hypothesis: That single dose oral dexamethasone 8mg reduces the proportion of patients who suffer rebound headache after treatment for migraine in the ED.

DETAILED DESCRIPTION:
Migraine headache can be a debilitating condition. A small but significant proportion of sufferers seek treatment in emergency departments [ED], accounting for 2-5% of ED visits.Available data suggests that up to 66% of these patients may experience rebound headache after discharge that affects their ability to function normally [eg work, social, etc].It appears that inflammation plays a key role in recurrences. A number of small studies suggest that a single dose of corticosteroids at the time of discharge might prevent rebound headache. To date these studies have used intravenous dexamethasone. The aim of this project is to determine if a single dose of oral dexamethasone at the time of discharge from the ED [after successful treatment] prevents rebound headache.

Hypothesis: That single dose oral dexamethasone 8mg reduces the proportion of patients who suffer rebound headache after treatment for migraine in the ED.

Aims: The primary aim is to compare the proportion of patients who experience rebound headache within 48 hours after ED treatment of migraine between a group treated with single dose oral dexamethasone 8mg and a group treated with placebo. Secondary aims are to compare headache severity, analgesia/ health service use, adverse events and return to normal functioning between the groups.

Methods:

Study design: Double blind, randomised placebo controlled clinical trial. Setting: Emergency Department, Western Hospital. Participants: Adult patients [age >17 years] with physician-diagnosed migraine treated in the ED.

Inclusion criteria: Consenting adult patients [age >17 years] with physician-diagnosed migraine treated in the ED who are willing and able to be contacted between 48-72 hours after discharge for follow-up.

Sample size: 76 patients. Note: The study was stopped early for operational reasons. 63 patients were analysed.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult patients [age >17 years] with physician-diagnosed migraine treated in the ED who are willing and able to be contacted between 48-72 hours after discharge for follow-up

Exclusion Criteria:

* Failure to consent
* Pregnancy
* Allergy to study medication
* Findings inconsistent with migraine
* Patients requiring hospital admission for further investigation and treatment
* Patients with active peptic ulcer disease
* Patients with Type 1 diabetes
* Patients taking corticosteroids for another condition within 7 days
* Active systemic fungal infection
* Patients previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-04; Primary Completion 2006-12 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Maree Kelly, MB BS, Principal Investigator — The Joseph Epstein Centre for Emergency Medicine Research
Locations (1):
- Department of Emergency Medicine, Western Health, Melbourne, Victoria, Australia

REFERENCES:
- [Result] Kelly AM, Kerr D, Clooney M. Impact of oral dexamethasone versus placebo after ED treatment of migraine with phenothiazines on the rate of recurrent headache: a randomised controlled trial. Emerg Med J. 2008 Jan;25(1):26-9. doi: 10.1136/emj.2007.052068. PMID 18156535

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Dexamethasone
Started | 32 | 31
Completed | 31 | 30
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dexamethasone | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 31 | 63
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13) | 37 (11) | 39 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  Australia | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Were Discharged Pain Free That Have a Recurrence of Headache Within 48 Hours.
Description: Proportion of patients who were discharged pain free who report recurrence of headache within 48 hours, on telephone followup.
Time Frame: 48 hours
Measure: Number; unit: Participants
Arm/Group | Placebo | Dexamethasone
Number analyzed (Participants) | 31 | 30
Participants | 13 | 14

2. Primary Outcome: Proportion of Patients With Recurrent Headache Within 48 Hours.
Description: Proportion of patients who report recurrent headache within 48 hours, on telephone followup.
Time Frame: 48 hours
Measure: Number; unit: Partcipants
Arm/Group | Placebo | Dexamethasone
Number analyzed (Participants) | 31 | 30
Partcipants | 12 | 8

3. Secondary Outcome: Proportion of Patients Requiring Additional Analgesia Within 48 Hours for Headache.
Description: Proportion of patients reporting a requirement for additional analgesia within 48 hours of treatment for headache, by telephone followup.
Time Frame: 48 hours
Measure: Number; unit: Participants
Arm/Group | Placebo | Dexamethasone
Number analyzed (Participants) | 31 | 30
Participants | 19 | 18

4. Post Hoc Outcome: Proportion of Patients With Recurrent Headache Within 48 Hours for Patient Subgroup With Duration of Migraine Less Than 24 Hours
Description: Proportion of patients who report recurrent headache within 48 hours for the patient subgroup with duration of migraine less than 24 hours
Time Frame: 48 hours
Measure: Number; unit: Participants
Arm/Group | Placebo | Dexamethasone
Number analyzed (Participants) | 21 | 20
Participants | 9 | 3

ADVERSE EVENTS:
Arm/Group | Placebo | Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 7/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Dexamethasone (N=31)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
flushing (Vascular disorders) | 0 (0) | 2 (2)
tingling (Nervous system disorders) | 0 (0) | 2 (2) — transient tingling in arms or feet
blurred vision (Eye disorders) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No